CLINICAL TRIAL: NCT06582693
Title: Refer2Quit: Evaluating a Proactive, Tailored, Population Health Approach for Tobacco Treatment for Household Smokers Through a Pediatric Care Network
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-021075; 1R37CA282153-01 (NIH)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Smoking; Smoking Cessation; Second Hand Tobacco Smoke
Keywords: Smoking; Smoking Cessation; Second Hand Tobacco Smoke
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Only adult participants will be blinded during the study. Child participants do not need to be blinded because they will not be engaging in study procedures. Study staff will be aware of the assigned treatment arms. To maintain the blinding of adult participants, study staff will not disclose the treatment assignment to the adult participants at any point during the study. The recruit and consent procedures will describe the study, but not provide the adult participants with details that would reveal their treatment assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Adult intervention arm participants will receive motivational counseling provided by the study staff member enrolling them. The study team member will offer 4 evidence-based treatment options (varenicline, NRT, quitline, and/or smokefreeTXT), emphasizing that the combination is often more effective than one treatment alone, and that they could start treatment even if they are not ready to quit.
  Interventions: Other: Refer2Quit
- Control Arm (No Intervention): Adult control arm participants will receive a handout listing tobacco treatment options that they can connect to on their own

INTERVENTIONS:
Other: Refer2Quit — The Refer2Quit intervention consists of automatic connection to the adult participant's choice of any or all of four evidence-based tobacco treatment options (varenicline, NRT, quitline, and/or smokefreeTXT), as well as motivational counseling provided by the study team. Supportive and motivational text messaging is also included in the intervention to connect or reconnect adult participants to treatments as needed. Text messaging and support would also focus on supporting appropriate use of NRT and/or varenicline if indicated.
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to compare the reach and effectiveness of the Refer2Quit intervention for increasing tobacco use treatment and quit rates among household members who smoke versus a treatment as usual group. This clinical trial also aims to study household member and pediatric patient characteristics that are associated with reach and effectiveness of Refer2Quit.

DETAILED DESCRIPTION:
This study aims to evaluate a proactive and population health-based approach that leverages a clinical decision support (CDS) system embedded in the electronic health record (EHR) to identify household members who smoke but did not complete the smoking survey at the visit, and remotely engage them in tobacco use treatment.

Participants will be recruited through up to 32 outpatient primary care practice from the Children's Hospital of Philadelphia's (CHOP) Pediatric Research Consortium (PeRC). Potential participants will be identified from the cohort of referrals for tobacco cessation treatment. Randomization of adult participants into either the intervention or control group will occur after the participants have consented to partake in the study and completed enrollment. The investigators will deploy a remote recruitment strategy (via phone and/or text) to outreach to eligible adult participants to maximize recruitment efforts.

After the initial referral of the household member who smokes, a study team member will reach out to them, explain the reason they are being contacted and confirm their smoking status and age. All participants will complete the enrollment step with data collection including: adult participant demographics, nicotine dependence and quitting motivation.

Only the intervention arm will receive the opportunity to be automatically connected by the study team to four evidence-based tobacco treatment options: varenicline, nicotine replacement therapy (NRT), quitline, and/or smokefreeTXT. Adult intervention arm participants will also receive brief motivational counseling by the study team.

Adult control arm participants will receive treatment as usual which consistent of a handout of evidence tobacco treatment resources which the adult participant must connect with on their own

Enrolled adult participants in both the intervention and control arms will be followed-up via surveys at approximately 1 and 6-month time intervals. Adult participants who self-report 7-day abstinence at the 1 and 6-month surveys will be asked to confirm smoking cessation through carbon monoxide testing.

ELIGIBILITY:
Adult Intervention Subject Inclusion Criteria

* Males or females ages ≥18 years in age
* Self-identify as a current combustible tobacco user
* Have a valid cell phone number

Child Intervention Subject Inclusion Criteria

* Must be a CHOP patient

Adult Intervention Subject Exclusion Criteria

* <18 years in age.
* Indicates no combustible tobacco smoking

Child Intervention Subject Exclusion Criteria

* Not a CHOP patient

Adult Control Subject Inclusion Criteria

* Males or females ages ≥18 years in age
* Self-identify as a current combustible tobacco user
* Have a valid cell phone number

Child Control Subject Inclusion Criteria

* Must be a CHOP patient

Adult Control Subject Exclusion Criteria

* <18 years in age.
* Indicates no combustible tobacco smoking

Child Control Subject Exclusion Criteria

* Not a CHOP patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of adult participants who engage in any evidence-based tobacco use treatments | Baseline, 1 and 6 months
  The proportion of adult participants who engage in any evidence-based tobacco use treatments, between the intervention and control arms, by adult participant self-report.
Combustible tobacco quit rate at 1 and 6 months | 1 and 6 months
  The quit rate, compared between the intervention and control arms, will be assessed by a self-reported 7-day point prevalence smoking abstinence, collected via follow-up survey, and confirmed via breath carbon monoxide (CO) <5ppm at the time-point

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Jenssen, MD, MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
For adult participants who sign up for the Quitline, the generated reports that contain participant names and contact information will be stored on a secure HIPAA-compliant server managed by CHOP. The reports will contain adult participants' identifiable information (e.g., name, phone number).
  For adult participants who sign up for SmokefreeTXT, their contact information and preference to enroll into the SmokefreeTXT program will be stored on a secure HIPAA-compliant server managed by CHOP. These reports will contain adult participants' identifiable information (e.g., name, phone number).
  For adult participants who sign up for varenicline and/or NRT, their contact information and preference to get the varenicline and/or NRT medication will be stored on a secure HIPAA-compliant server managed by CHOP. These reports will contain adult participants' identifiable information (e.g., name, phone number).
Supporting Information: Study Protocol
Time Frame: Data will be shared with key stakeholders throughout the duration of the study.
Access Criteria: Data will be restricted to appropriately authorized members of the study team.